CLINICAL TRIAL: NCT03273322
Title: Assessment of Dual Antiplatelet Therapy Versus Rivaroxaban In Atrial Fibrillation Patients Treated With Left Atrial Appendage Closure: The Randomized ADRIFT Study
Brief Title: Assessment of Dual Antiplatelet Therapy Versus Rivaroxaban In Atrial Fibrillation Patients Treated With Left Atrial Appendage Closure
Acronym: ADRIFT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Action Research Group (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P161102J
Record Dates: First submitted 2017-08-11; First posted 2017-09-06 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Atrial Fibrillation; Atrial Appendage; Hemorrhage
Keywords: Left atrial appendage closure; Rivaroxaban; Dual antiplatelet therapy; Anticoagulation; Stroke prevention
MeSH Terms: conditions — Atrial Fibrillation; Hemorrhage | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1: Rivaroxaban 10 mg qd (Experimental): Rivaroxaban 10 mg, 1 tablet a day, from randomization to Day 90 should be taken between 8 and 10 AM
  Interventions: Drug: Rivaroxaban 10 mg qd
- 2: Rivaroxaban 15 mg qd (Experimental): Rivaroxaban 15 mg, 1 tablet a day, from randomization to Day 90
  should be taken between 8 and 10 AM
  Interventions: Drug: Rivaroxaban 15 mg qd
- 3: DAPT (Active Comparator): Aspirin 75 mg, 1 a day Clopidogrel 75 mg, 1 tablet a day from randomization to Day 90 should be taken between 8 and 10 AM
  Interventions: Drug: DAPT

INTERVENTIONS:
Drug: Rivaroxaban 10 mg qd — 10mg qd
  Other Names: Experimental
  Arms: 1: Rivaroxaban 10 mg qd
Drug: Rivaroxaban 15 mg qd — 15mg qd
  Other Names: Experimental
  Arms: 2: Rivaroxaban 15 mg qd
Drug: DAPT — Aspirin 75 mg qd + Clopidogrel 75 mg qd
  Other Names: Active comparator
  Arms: 3: DAPT

SUMMARY:
Evaluation of 2 doses of rivaroxaban (10 and 15 mg) compared to dual anti platelet therapy (aspirin+clopidogrel) after left atrial appendage closure. The patients will be assessed at 10 and 90 days: central laboratory hemostasis analysis and clinical events assessment.

DETAILED DESCRIPTION:
Data on antithrombotic therapy after Left Atrial Appendage Closure (LAAC) are scarce and no randomized evaluation has been performed to demonstrate what is the best antithrombotic strategy following LAAC. LAAC is classically associated with a 6-week period of anticoagulation with warfarin + aspirin followed by once daily clopidogrel (75 mg) + aspirin (81-325 mg) until the 6 months visit, then aspirin alone is continued indefinitely, as tested in patients without contraindication for anticoagulation in the pivotal Watchman trials. LAAC is mostly used in Europe as an alternative to warfarin anticoagulation when patients have a contraindication to or are unsuitable for warfarin anticoagulation. The classic regimen is not applicable and believed to be too risky in such frail patients. These patients usually receive a regimen of daily clopidogrel + aspirin followed by single antiplatelet therapy (most frequently used treatment). Some patients receive oral anticoagulation without aspirin, including NOAC anticoagulation. Rivaroxaban is a tempting strategy for anticoagulation following LAAC in atrial fibrillation (AF) patients. The dose needs first to be carefully evaluated the trial propose a dose ranging study in patients who have undergone successful LAAC.

The study will evaluate two different Rivaroxaban regimen (10 or 15 mg a day) in comparison to dual antiplatelet therapy (DAPT) (aspirin+clopidogrel : control arm representing standard of care) after successful LAAC. The aim is to investigate whether rivaroxaban could provide correct anticoagulation levels and adequately suppress coagulation activation after LAAC.

The patient will be enrolled after left atrial appendage closure before discharge. The randomization is 1/1/1 between the 3 groups : rivaroxaban 10mg a day, rivaroxaban 15 mg a day and aspirin 75mg + clopidogrel 75 mg a day. At 10 and 90 days, the patients will be sampled for biological assessment : Prothrombin fragments 1+2, Factor Xa inhibitory activity, Russel Viper venom enzyme assay, thrombin anti-thrombin (TAT) complex, D-Dimers, Prothrombin time (Neoplastin) and plasma von Willebrand factor (vWf) Ag level

After 90 days, the patient will end his/her participation in the trial. Clinical endpoints (death, MI, Stroke, TIA, systemic embolism, extracranial major bleeding or clinically relevant non major bleeding) at 90 days will be assessed by a clinical endpoint committee. Central echographic laboratory will review all 90 days transesophageal echocardiography (TEE) to detect the presence of thrombus or peri-device leak.

The study is open-label. Central laboratory, clinical endpoint committee and echographic core laboratory is blinded to randomization arm.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age
* Patients who underwent a clinically successful LAAC procedure (device implanted without procedural or bleeding complication). LAAC may have been indicated for patients contraindicated or unsuitable for long-term Vitamin K antagonists (VKA) anticoagulation.
* AF (permanent or persistent or paroxysmal) patients irrespective of prior antithrombotic treatment are eligible for randomization.
* Written informed consent by the patient or designee if the patient is unable to consent
* Patients affiliated to the French social security system

Exclusion Criteria:

* Creatinine clearance <30 mL / min (Cockcroft formula).
* Dialysis.
* Mechanical heart valves or valvular disease requiring surgery or interventional procedure
* Planned Ablation of AF during follow up period
* Mandatory indication for dual antiplatelet therapy (e.g. recent stent) or single anti-platelet treatment (SAPT) (e.g. high coronary risk).
* Any contra-indication or known allergy to aspirin or clopidogrel or rivaroxaban.
* Any mandatory indication for anticoagulation for a reason other than AF (e.g. Pulmonary embolism)
* Ongoing major bleeding or complicated or recent (<72hours) major surgery
* Known large oesophageal varices or decompensated liver disease (unless a documented positive opinion of a gastro-enterologist)
* Severe thrombocytopenia (<50,000/ml) after referral to haematologist to confirm or not contraindication
* Recent myocardial infarction (<6 weeks).
* Recent cerebro-vascular event (CVE) or transient ischemic attack (<6 weeks) after evaluation of stroke vs bleeding risk by the referring neurologist.
* Recent Intracranial bleeding (< 6 months): these patients will be evaluated by a neurologist as these patients may be considered at higher stroke risk. Neurologist may consider that the LAAC procedure with a short (90 days) period of anticoagulation or antiplatelet therapy as tested in the protocol is a preferable option (in that case intracranial hemorrhage (ICH) will not be considered as a contraindication).
* Prasugrel or ticagrelor concomitant use
* Participating in an investigational drug or another device trial within the previous 30 days.
* High likelihood of being unavailable for follow-up or psycho-social condition making study participation impractical.
* Woman with child bearing potential who do not use an efficient method of contraception.
* positive serum or urine pregnancy test for woman with child bearing potential
* Pregnancy or within 48 hours post-partum or breast feeding women
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Measure of prothrombin fragment 1 + 2 | at Day 10
  Measure of prothrombin fragment 1 + 2 at Day 10 (2 to 4 hours after last intake : concentration peak)

SECONDARY OUTCOMES:
Measure of prothrombin fragment 1 + 2 | at Day 90
  Measure of prothrombin fragment 1 + 2 at Day 90 (2 to 4 hours after last intake : concentration peak)
Factor Xa inhibitory activity at day 10 | at Day 10
  Factor Xa inhibitory activity
Factor Xa inhibitory activity at day 90 | at Day 90
  Factor Xa inhibitory activity
Russel Viper venom enzyme assay | at Day 90
  Russel Viper venom enzyme assay
TAT complex | at Day 10
  TAT complex
TAT complex | at Day 90
  TAT complex
D-Dimers | at Day 10
  D-Dimersand at peak, 2 to 4 hours after treatment intake
D-Dimers | at Day 90
  D-Dimersand at peak, 2 to 4 hours after treatment intake
Prothrombin time (Neoplastin) | at Day 10
  Prothrombin time (Neoplastin)
Prothrombin time (Neoplastin) | at Day 90
  Prothrombin time (Neoplastin)
Plasma vWf Ag level | at Day 10
  plasma vWf Ag level treatment intake
Plasma vWf Ag level | at Day 90
  plasma vWf Ag level treatment intake
Haemorrhagic stroke and bleeding will be safety outcomes TEE with central core lab reading: presence of thrombus, peri-device leak | at Day 90
  Haemorrhagic stroke and bleeding will be safety outcomes 3-month TEE with central core lab reading: presence of thrombus, peri-device leak
Composite clinical endpoint combining all clinical outcomes | at Day 90
  Composite clinical endpoint combining all clinical outcomes : Death, MI, stroke, TIA,
Death (any cause) | at Day 90
  Death (any cause) assessed individually and combined at other outcomes
Myocardial infarction (MI) | at Day 90
  Myocardial infarction (MI) assessed individually and combined at other outcomes
Stroke (ischaemic stroke, haemorrhagic stroke) | at Day 90
  Stroke (ischaemic stroke, haemorrhagic stroke) assessed individually and combined at other outcomes
Transient Ischemic Attack (TIA) | at Day 90
  Transient Ischemic Attack (TIA) assessed individually and combined at other outcomes
Systemic embolism | at Day 90
  Systemic embolism assessed individually and combined at other outcomes
Extracranial major bleeding or clinically relevant non major bleeding (ISTH definition) at day 90 | at Day 90
  Extracranial major bleeding or clinically relevant non major bleeding (ISTH definition) assessed individually and combined at other outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Gilles MONTALESCOT, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Pitié-Salpêtrière Paris
Locations (1):
- Institut de Cardiologie - Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duthoit G, Silvain J, Marijon E, Ducrocq G, Lepillier A, Frere C, Dimby SF, Popovic B, Lellouche N, Martin-Toutain I, Spaulding C, Brochet E, Attias D, Mansourati J, Lorgis L, Klug D, Zannad N, Hauguel-Moreau M, Braik N, Deltour S, Ceccaldi A, Wang H, Hammoudi N, Brugier D, Vicaut E, Juliard JM, Montalescot G. Reduced Rivaroxaban Dose Versus Dual Antiplatelet Therapy After Left Atrial Appendage Closure: ADRIFT a Randomized Pilot Study. Circ Cardiovasc Interv. 2020 Jul;13(7):e008481. doi: 10.1161/CIRCINTERVENTIONS.119.008481. Epub 2020 Jul 17. PMID 32674675